CLINICAL TRIAL: NCT04200144
Title: An Open-label, Randomized, Controlled Clinical Trial on the Effects of Endoscopic Sleeve Gastroplasty on Weight, Metabolic Risk Factors, Quality of Life, Satiety, Gastrointestinal Motility and Gut Microbiota
Brief Title: Endoscopic Sleeve Gastroplasty for Obesity and Microbiota Randomized Trial
Acronym: ESGORT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, BOSKOSKI IVO, MD, PhD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2837
Record Dates: First submitted 2019-11-14; First posted 2019-12-16 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Obesity; Endoscopic Sleeve Gastroplasty; Gastric Motility; Gastric Hormones; Microbiota; Quality of Life
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active endoscopic treatment (Active Comparator): Patients that will undergo Endoscopic Sleeve Gastroplasty
  Interventions: Device: Endoscopic sleeve gastroplasty
- standard medical therapy control diet group (Active Comparator): Patients that will undergo diet
  Interventions: Device: Endoscopic sleeve gastroplasty

INTERVENTIONS:
Device: Endoscopic sleeve gastroplasty — Endoscopic sleeve gastroplasty with Overstitch (Apollo Endosurgery)

SUMMARY:
This is an interventional, open-label, randomized (2:1), standard medical therapy-controlled trial.

Subjects in the standard therapy group will be given the opportunity to undergo the active endoscopic treatment after 6 months of follow up (open label extension) if they will not achieve an adequate result on body weight. All patients will be followed until the planned end of the study after 36 months from the ESG procedure.

To study the effects of endoscopic gastroplasty on weight, metabolic risk factors, quality of life, satiety, gastrointestinal motility and gut microbiota compared to standard medical treatment control group.

Primary endpoint:

- Total body weight loss (%)

Secondary endpoints:

* Metabolic risk factors (e.g. lipid profile) and anthropometric measurements (e.g hip and waist circumference)
* Body composition
* Quality of life
* Gastroesophageal reflux disease
* Non-Alcoholic Fatty Liver Disease (NAFLD)
* Non- Alcoholic-Steato-Hepatitis (NASH)
* Satiety
* Gut microbiota

Exploratory endpoints:

* Gut hormones e.g. glucagon-like peptide 1, PYY and ghrelin
* Gastrointestinal motility

ELIGIBILITY:
Inclusion Criteria:

The participants have to fulfill the following criteria for participating in the study:

* Age 20 to 65 years
* BMI between 30 to 45 kg/m2
* Willingness to participate in the study and ability to comply and understand the study protocol

Exclusion Criteria:

Active gastric ulcer during the last 6 months

* Organic or motility disorder of the stomach and / or esophagus
* Anticoagulant treatment
* Previous bariatric surgery or any other type of surgery of the esophagus, stomach and duodenum
* Ongoing or active malignancy during the last 5 years
* Myocardial infarction during the past 6 months or/and heart failure class III or IV according to the New York Heart association's classification
* Drug or alcohol abuse
* Bulimic or binge eating pattern
* Continuous glucocorticoid or anti-inflammatory treatment
* Uncontrolled thyroid disease
* Pregnancy, breastfeeding
* Psychiatric or cooperative problems or low compliance that is a contraindication from participating in the study
* Hiatal hernia > 5 cm
* Currently participating in other study
* Any health issue that might put the patient at risk if the treatment is performed, judged by the investigator

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-02-04 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2025-12-02 (Estimated)

PRIMARY OUTCOMES:
Total body weight loss | 12 months
  Total body weight loss (%) measurement in kg and BMI
Total body weight loss | 36 months
  Total body weight loss (%) measurement in kg and BMI

SECONDARY OUTCOMES:
Non-Alcoholic Fatty Liver Disease evaluation | 12 months
  Non-Alcoholic Fatty Liver Disease
Non- Alcoholic-Steato-Hepatitis evaluation | 12 months
  Non- Alcoholic-Steato-Hepatitis
Gut microbiota characterization | 6 months
  Gut microbiota
Evaluation for Gastroesophageal reflux disease | 12, 24, 36 months
  Gastroesophageal reflux disease
Gut hormones e.g. glucagon-like peptide 1, PYY and ghrelin dosages | Baseline and 6 months
  Gut hormones e.g. glucagon-like peptide 1, PYY and ghrelin
performing of gastric emptying scintigraphy for gastrointestinal motility | Baseline and six months
  Gastrointestinal motility evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided